CLINICAL TRIAL: NCT02837380
Title: An Open Label Study to Evaluate the Pharmacokinetics of Fluticasone Furoate /Umeclidinium Bromide/Vilanterol (100/62.5/25 mcg) After Single and Repeat Dose Administration From a Dry Powder Inhaler in Healthy Chinese Subjects
Brief Title: A Phase I Pharmacokinetic Study of Fluticasone Furoate /Umeclidinium Bromide/Vilanterol (100/62.5/25 Microgram [mcg]) After Single and Repeat Dose Administration From a Dry Powder Inhaler in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200558
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Long-acting muscarinic antagonist; Long-acting beta2 agonist; Dry powder inhaler; Inhaled corticosteroid
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FF/UMEC/VI (Experimental): Subjects will receive single combination dose of FF/UMEC/VI 100/62.5/25 mcg via a DPI in the morning for 7 days.
  Interventions: Drug: FF; Drug: VI/UMEC

INTERVENTIONS:
Drug: FF — FF is a dry white powder blended with lactose. It is the first strip of DPI. Per blister contains 100 mcg of dose
Drug: VI/UMEC — VI and UMEC bromide combination is a dry white powder blended with lactose and magnesium stearate. It is the second strip of DPI. Per blister contains 25 mcg/62.5 mcg of VI/UMEC dose

SUMMARY:
This is an open-label study to evaluate the PK of FF/UMEC/VI in dose combinations of 100/62.5/25 mcg after single and repeat dose administration from a DPI in healthy Chinese subjects. This study will evaluate the systemic pharmacokinetics (PK), of FF/UMEC/VI in Chinese healthy population when administered using dry powder inhaler (DPI)as a blended combination of UMEC/VI in one strip and FF in the second strip in dose combinations of 100/62.5/25 mcg. The triple, fixed dose combination product Fluticasone furoate(FF)/ Vilanterol (VI) /Umeclidinium bromide (UMEC) with new configuration enables the delivery of inhaled long-acting muscarinic antagonist (LAMA), Long-acting beta2 agonist (LABA) and inhaled corticosteroid (ICS) from a single device. Approximately 16 subjects will be enrolled in the study. After taking into account the allowable time windows for screening, treatment and follow-up, a subject will be in the study for a maximum duration of 6-7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* No significant abnormality on 12-lead ECG at screening, including the following specific requirements: Ventricular rate inside the range 40-90 beats (inclusive) per minute (bpm) at screening, PR interval <=210milliseconds (msec), No pathological Q waves, QRS interval >=60 msec and <=120 msec, the waveforms must enable the QT interval to be clearly defined and the corrected QT interval by Fridericia's method (QTcF) must be <450msec (machine or manual reading) based on a single ECG value, or an average from three ECGs obtained over a brief recording period.
* Forced Expiratory Volume in 1 second (FEV1) >=80% predicted and a FEV1/Forced Vital Capacity (FVC) ratio >=0.7
* AST, ALT, ALP and bilirubin <=1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Male/females aged between 18 and 45 years of age (inclusive), at the time of signing the informed consent. Male and female is 1:1.
* Body weight >=50 Kilogram (Kg) and Body Mass Index (BMI) within the range 19-24 Kg per square meter (m^2) (inclusive).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and lung function testing. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the investigator considers the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures and outcome.
* Subjects who are current non-smokers and have not used any tobacco products in the 6 month period preceding screening and have a pack history of <=10 pack years.

[Number of pack years = (number of cigarettes per day /20) x number of years smoked]

* Capable of giving written informed consent.
* A female subject is eligible to participate if: she is of child-bearing potential and is abstinent or agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the chance of pregnancy at that point or She must agree to use contraception until the follow-up visit (i.e. until follow-up visit is complete) or she is on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method or she is confirmed postmenopausal or permanently sterilised (example [e.g.] tubal occlusion, tubal ligation, hysterectomy, bilateral salpingectomy).

Exclusion Criteria:

* Lactating or pregnant females as determined by positive serum or urine human chorionic gonadotropin (HCG) test at screening or prior to dosing.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities or a history of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a 285 milliliter (mL) glass of full strength beer or 425 mL schooner of low strength beer or 1 (30 mL) measure of spirits or 1 glass (100 mL) of wine
* History of chronic respiratory problems (i.e. history of asthmatic symptoms) in the last 10 years or suffered an upper or lower respiratory tract infection within 4 weeks of the screening visit.
* A positive pre-study Hepatitis B surface antigen (HBsAg) or positive Hepatitis C antibody result within 3 months of screening or a positive test for Human Immunodeficiency Virus (HIV) antibody or Syphilis antibody.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator the medication will not interfere with the study procedures or compromise subject safety.
* A positive pre-study drug/alcohol screen or on admission to the Unit.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) or has had exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unwillingness or inability to follow the study procedures outlined in the protocol.
* The subject is unable to refrain from the consumption of red wine, seville oranges, grapefruit or grapefruit juice and pummelos, exotic citrus fruits, grapefruit hybrids or any fruit juices containing these fruits from 7 days prior to the first dose of study medication and for the duration of the study.
* Mentally or legally incapacitated.
* History of allergy or hypersensitivity to heparin, or any corticosteroid, anticholinergic/muscarinic receptor antagonist, beta-2 agonist, lactose/milk protein or magnesium stearate or a history of drug allergy or other allergy that, in the opinion of the investigator, contraindicates their participation.
* A chest X-ray or computed tomography (CT) scan that reveals evidence of clinically significant abnormalities. A chest X-ray must be taken before Day1, in any day between screening and Day -1(inclusive) if a chest X-ray or CT scan is not available within 6 months prior to screening day.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of FF, UMEC and VI after single inhaled dose on Day1 | Pre-dose, 5 minutes (min), 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 hour (h), 1.5 h, 2 h, 4 h, 6 h and 8 h post dose on Day 1
Time of occurrence of Cmax (tmax) of FF, UMEC and VI after single inhaled dose on Day1 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 hour (h), 1.5 h, 2 h, 4 h, 6 h and 8 h post dose on Day 1
Area under the concentration time curve (AUC) between zero and the time to the last measurable concentration (AUC (0-t)) of FF, UMEC and VI after single inhaled dose on Day1 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 hour (h), 1.5 h, 2 h, 4 h, 6 h and 8 h post dose on Day 1
AUC from time zero (pre-dose) to the time of last common measurable time-point within subject /treatment/study (AUC (0-t')) of FF, UMEC and VI after single inhaled dose on Day1 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 hour (h), 1.5 h, 2 h, 4 h, 6 h and 8 h post dose on Day 1
Elimination rate constant (kel) of FF, UMEC and VI after single inhaled dose on Day1 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 hour (h), 1.5 h, 2 h, 4 h, 6 h and 8 h post dose on Day 1
Terminal half-life (t1/2) of FF, UMEC and VI after single inhaled dose on Day1 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 hour (h), 1.5 h, 2 h, 4 h, 6 h and 8 h post dose on Day 1
AUC between zero and the infinity (AUC (0-inf)) of FF, UMEC and VI after single inhaled dose on Day1 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 hour (h), 1.5 h, 2 h, 4 h, 6 h and 8 h post dose on Day 1
tmax after repeat inhaled dose of FF, UMEC and VI on Day 7 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, and 24 h post dose on Day 7
AUC (0-t) of FF, UMEC and VI after repeat inhaled dose on Day 7 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, and 24 h post dose on Day 7
AUC (0-t') of FF, UMEC and VI after repeat inhaled dose on Day 7 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, and 24 h post dose on Day 7
Maximum concentration observed at steady state (Css_max) of FF, UMEC and VI after repeat inhaled dose on Day 7 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, and 24 h post dose on Day 7
Minimum concentration observed at steady state (Css_min) of FF, UMEC and VI after repeat inhaled dose on Day 7 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, and 24 h post dose on Day 7
Average steady state concentration (Css_av) of FF, UMEC and VI after repeat inhaled dose on Day 7 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, and 24 h post dose on Day 7
AUC at steady state (AUCss) of FF, UMEC and VI after repeat inhaled dose on Day 7 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, and 24 h post dose on Day 7
Observed accumulation ratio (Ro) of FF, UMEC and VI after repeat inhaled dose on Day 7 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, and 24 h post dose on Day 7
Maximum observed concentration ratio (RCmax) of FF, UMEC and VI after repeat inhaled dose on Day 7 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, and 24 h post dose on Day 7
Degree of fluctuation (DF) of FF, UMEC and VI after repeat inhaled dose on Day 7 | Pre-dose, 5 min, 8 min, 10 min, 12 min, 15 min, 30 min, 45 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h, 12 h, and 24 h post dose on Day 7

SECONDARY OUTCOMES:
Number of subjects with any Adverse Events (AEs) and any serious adverse events (SAEs) | Up to Day 17
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement and associated with liver injury and impaired liver function will be categorized as SAE.
Pulse rate as a measure of safety | Up to Day 17
  Pulse rate will be taken in sitting position having rested in this position for at least 5 minutes
Systolic and diastolic blood pressure as a measure of safety | Up to Day 17
  Systolic and diastolic blood pressure will be taken in sitting position having rested in this position for at least 5 minutes
Electrocardiogram (ECG) as a measure of safety | Up to Day 17
  12-Lead ECG will be taken in a supine position, having rested in this position for at least 5 minutes.
Number of subjects with abnormal hematology values | Up to Day 17
  Hematological parameters includes: platelet count, red blood cell (RBC) count, absolute white blood cell (WBC) count, hemoglobin, hematocrit, RBC indices (includes: mean corpuscular volume [MCV], mean corpuscular hemoglobin [MCH], MCH concentration [MCHC]) and WBC differential count (includes: neutrophils, lymphocytes, monocytes, eosinophils and basophils)
Number of subjects with abnormal clinical biochemistry values | Up to Day 17
  Clinical chemistry includes: blood Urea Nitrogen (BUN), creatinine, Glucose (fasting), potassium, chloride, calcium, sodium, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyltransferase (GGT), alkaline phosphatase (ALP), total and direct bilirubin, uric acid, albumin and total protein
Number of subjects with abnormal urinalysis results | Up to Day 17
  Urinalysis includes: Specific gravity, analysis of pH, glucose, protein, blood & ketones by dipstick method, and microscopic examination (if blood or protein is abnormal)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

REFERENCES:
- [Derived] Li Y, Li H, Sheng Y, Du X, Yao Y, Luo X, Ma P. Pharmacokinetics of Single and Repeat Doses of Fluticasone Furoate/Umeclidinium/Vilanterol in Healthy Chinese Adults. Clin Pharmacol Drug Dev. 2019 Aug;8(6):721-733. doi: 10.1002/cpdd.626. Epub 2018 Nov 14. PMID 30427594